CLINICAL TRIAL: NCT00486590
Title: The Evaluation of Prolact-Plus, Human Milk Fortifier (Human, Pasteurized) for Pre-term Infants Receiving Human Milk
Brief Title: Evaluation of Prolact-Plus Human Milk Fortifier
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prolacta Bioscience (Industry)
Responsible Party: Martin L. Lee, PhD; Chief Scientific Officer, Prolacta Bioscience
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MPPF 001-2006
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2008-02

CONDITIONS: Infant, Very Low Birth Weight
Keywords: Human milk fortification; Premature neonate; Very low birth weight
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Prolact-Plus Human Milk Fortifier

SUMMARY:
Prolacta Bioscience has developed the first purely human fortifier, Prolact-Plus, that can provide a source of many of the required nutrients for premature, newborn infants, particularly protein and calories. This product is made from donor human milk from which the skim (non-lipid portion) has been separated and then concentrated. A certain amount of the lipid content has been added back to achieve higher caloric content within a small delivery volume. The product is then pasteurized and filled in small quantities in order to allow for the addition of mother's own milk (or, possibly, milk from another donor). The goal of the preparation is to achieve an increase of approximately 4 cal/oz of mother's milk and to provide a protein level (when mixed with average pre-term milk) of about 3.5-3.8 g/100 Kcal of feed.

The data on Prolact-Plus will be obtained prospectively from infants who will receive human milk fortified in this fashion. The data on standard,bovine (cow)-fortified milk will be obtained retrospectively from medical records at the participating institutions. While this design is not necessarily optimal in this setting, it is an efficient and quick approach to evaluating the acute clinical effect of Prolact-Plus. It is anticipated that further studies will be conducted that will examine longer-term accounts and possibly do this in a controlled, randomized environment.

The goal of this study is to evaluate the short-term effect of Prolact-Plus fortified human milk when compared with bovine-based fortification of human milk on parameters such as growth and short-term development, infectious complications and incidence of feeding intolerance in a cohort design. Statistically, the study will attempt to evaluate a null hypothesis of equivalent results with respect to these parameters between the two types of fortifiers as compared with a two-sided alternative (difference between the groups).

In addition, data will be collected on overall survival and length of stay in the NICU. These data will be collected for descriptive purposes, although an attempt will be made to compare the findings with those obtained from the bovine-based fortifier.

DETAILED DESCRIPTION:
This will be a cohort designed study in pre-term infants (<32 weeks of gestation) comparing bovine fortified (using any one of the commercially available fortifier products) human milk with Prolact-Plus (human) fortified human milk in which the former cohort will be obtained retrospectively and the latter obtained prospectively in each participating institution. The number of infants to be included in this study is a minimum of 50 in each group who complete the 30 days on study. (If a baby drops out of the study prior to 30 days of evaluation, then they would be replaced in order to achieve that number.) This sample size was not determined statistically, but rather is based solely on the desire to obtain a reasonable amount of data to evaluate the new human fortifier in this setting. However, from the perspective of a non-inferiority evaluation of an endpoint such as feeding intolerance, consider the following. Assuming a rate of 15% for this outcome for the retrospective cohort, then with 50 subjects per cohort, the study would be able to demonstrate a lack of inferiority of the human-based fortifier with a delta of 20% using a power of slightly greater than 80% and a one-sided 2.5% significance level. (By a "delta of 20%" it is implied that a theoretical feeding intolerance rate for the Prolact-Plus of no worse than 35% would result in a conclusion of lack of inferiority with the given levels of significance and power.) Conversely, if the human-based fortifier is able to reduce the feeding intolerance rate from 15% to about 1%, then with the sample sizes in this trial, this would be doable with 80% power and 5% significance (two-sided). (Thus, the trial, in theory, also could demonstrate a dramatic reduction in this rate.) The retrospective data will be obtained from available medical charts at the participating institution and the selected infants should reflect the most recently treated (within the 12 month period prior to the initiation of the prospective phase of this protocol) and the numbers should be similar in kind to the number treated prospectively in that institution.

ELIGIBILITY:
Inclusion Criteria:

1. Between 23 and 32 weeks gestational age
2. Weigh between 500 and 1600g
3. In the retrospective group, an infant must have been able to adhere to a feeding protocol that included only mother's own milk fortified by either bovine or human product from the time that enteral feeding began (or whenever fortified human milk feeding began) through the next 30 days of life or hospital discharge, whichever came first.
4. In the prospective group, the infant must be expected to be able to adhere to a feeding protocol that includes only mother's own milk fortified by the human product from the time that enteral feeding began (or whenever fortified human milk feeding began) through the next 30 days of life or hospital discharge, whichever comes first.
5. Informed consent obtained from parent or legal guardian.
6. Mother must be willing to adhere to a feeding protocol that includes 30 days of mother's own milk for the prospective arm of the study.

Exclusion Criteria:

1. Less than a 50% probability of survival through the study period (first 30 days of enteral feeding or hospital discharge).
2. On any other clinical study during the study period
3. Receipt of any bovine-based formula or fortifier prior to the infant's enrollment in the study.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2006-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Feeding intolerance | 30 days
Necrotizing enterocolitis | 30 days

SECONDARY OUTCOMES:
Length of stay in NICU and hospital | Indeterminate
Growth parameters, e.g. weight, head circumference, and length | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Martin L Lee, PhD, Study Director — Prolacta Bioscience
Locations (4):
- United States (4):
  - Shands Children's Hospital, Gainesville, Florida
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Miami Children's Hospital, Miami, Florida
  - Memorial Hospital of South Bend, South Bend, Indiana